CLINICAL TRIAL: NCT05382247
Title: Ultrasonographic Assessement Of Diaphragm In Neuromuscular Diseases In Pediatric Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Lamiaa Kamel Morssi, resident doctor at pediatric department ,faculty of medicine,sohag university, Sohag University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: Soh-Med-22-5-08
Record Dates: First submitted 2022-05-15; First posted 2022-05-19 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Ultrasonographic Assessement Of Diaphragm In Neuromuscular Diseases In Pediatric Patients
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pediatric patients with neuromuscular diseases (Active Comparator)
  Interventions: Device: ultrasonography
- children not suffering from neuromuscular diseases (Active Comparator)
  Interventions: Device: ultrasonography

INTERVENTIONS:
Device: ultrasonography — Full history taking, thorough clinical examination, review of participants medical files.
  Patients will be typically examined during spontaneous respiration to help assessement of diaphragmatic motion.
  The supine position will be used whenever possible to avoid overall variability, side-to-side variability, and for greater reproducibility.
  Patients can be examined in quiet respiration and during deep breathing or sniff maneuver.
  For uncooperative patients appropriate sedative for age will be used. Assessement of diaphragmatic function: the analysis of the dome excursion with M mode approach Evaluation of diaphragmatic thickness and thickening during inspiration by analyzing the apposition zone.

SUMMARY:
The diaphragm is the main muscle of respiration during resting breathing (1), and is formed by two muscles with dual innervation, joined by a central tendon. When it is contracted, the caudal movement increases the volume of the rib cage, generating the negative pressure necessary for inspiratory flow (2). When respiratory demands are increased or diaphragm function is impaired, rib cage muscles and expiratory muscles are progressively recruited. In some patients with diaphragm dysfunction, this compensation is associated with minimal or no respiratory symptoms. In other patients, this compensation is associated with significant respiratory symptoms. Early diagnosis of diaphragmatic dysfunction is essential, because it may be responsive to therapeutic intervention (3). The ultimate causes of diaphragmatic dysfunction can be broadly grouped into three major categories: disorders of central nervous system or peripheral neurons, disorders of the neuromuscular junction and disorders of the contractile machinery of the diaphragm itself (4). So In summary, motion and contractile force of the diaphragm may be affected by pathological alterations of the following anatomical structures:

* - Central nervous system
* - Phrenic nerve
* - Neuromuscular junction
* - Diaphragm muscle
* - Thoracic cage
* - Upper abdomen In patients on mechanical ventilation, the positive end expiratory pressure (PEEP) level also decrease diaphragmatic motion by increasing the end expiratory lung volume and thereby lowering the diaphragmatic dome at the end of expiration (3).

Diaphragm muscle dysfunction is increasingly recognized as an important element of several diseases including neuromuscular diseases leading to a restrictive respiratory pattern (1). The assessment of respiratory muscle function is of paramount interest in patients with neuromuscular disorders. In patients with neuromuscular diseases, respiratory symptoms are subtle and usually appear late in the clinical course of the disease, partly because of the limited mobility of patients due to peripheral muscle weakness, except in the case of acute respiratory failure due to infection. Clinical presentation is quite variable in cases of diaphragmatic failure. Orthopnea may be present and paradoxical abdominal motion may be observed during inspiration, with the abdomen moving inward while the rib cage expands (3). Different structural and functional techniques are available for evaluating the diaphragm. Each technique has its strengths and weaknesses (5). Imaging of respiratory muscles was divided into static and dynamic techniques. Static techniques comprise chest radiography, B-mode (brightness mode) ultrasound, CT and MRI, and are used to assess the position and thickness of the diaphragm and the other respiratory muscles. Dynamic techniques include fluoroscopy, M-mode (motion mode) ultrasound and MRI, used to assess diaphragm motion in one or more directions (6). The recent development of diaphragmatic ultrasound has revolutionized diaphragm evaluation (2). Diaphragm ultrasonography was first described in the late 1960s as a means to determine position and size of supra- and subphrenic mass lesions, and to assess the motion and contour of the diaphragm (1). Two decades later, Wait et al, developed a technique to measure diaphragm thickness based on ultrasonography. Later on the investigators reported a close correlation between diaphragm thickness measured in cadavers using ultrasound imaging and thickness measured with a ruler (7). it has been shown to be similar in accuracy to most other imaging modalities for diaphragm assessment (5), as it can be used to assess bilateral diaphragmatic morphology and function in real time, permitting follow-up without exposure to radiation. It is, moreover, affordable and ubiquitous. (2). First developed in intensive care, mainly for weaning from mechanical ventilation, its use is now extending to pulmonology. Different measurements are described such as diaphragmatic excursion, diaphragmatic thickness and diaphragmatic thickening fraction (8). US measurements of diaphragm muscle thickness and thickening with inspiration have been shown to be superior to phrenic nerve conduction studies (NCS), chest radiographs, and fluoroscopy for detection of neuromuscular disease affecting the diaphragm. The main use in pulmonology is for the respiratory evaluation of patients with neuromuscular diseases, for the search of isolated diaphragmatic impairment and for patients with chronic obstructive lung diseases. Numerous studies are in progress to better determine the role of diaphragmatic ultrasound (5).

ELIGIBILITY:
Inclusion Criteria:

Children and adolescents aged 6 months - 14 years, diagnosed with neuromuscular diseases, attending the Pediatric neurology clinic at Sohag University Hospital.

Exclusion Criteria:

* History of abdominal or thoracic surgery that may influence diaphragm motion.
* Prolonged mechanical ventilation as it may affect diaphragm thickness and motion.
* Presence of supra or subdiaphragmatic lesion limiting diaphragm motion

Ages: 6 Months to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2022-05-13 (Actual); Primary Completion 2023-05-13 (Estimated); Study Completion 2023-05-13 (Estimated)

PRIMARY OUTCOMES:
diaphragmatic excursion | 1 year
  To assess the diaphragmatic motion by M-mode

SECONDARY OUTCOMES:
diaphragmatic thickness | 1 year
  diaphragmatic thickness

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Laghi FA Jr, Saad M, Shaikh H. Ultrasound and non-ultrasound imaging techniques in the assessment of diaphragmatic dysfunction. BMC Pulm Med. 2021 Mar 15;21(1):85. doi: 10.1186/s12890-021-01441-6. PMID 33722215
- [Background] Sayas Catalan J, Hernandez-Voth A, Villena Garrido MV. Diaphragmatic Ultrasound: An Innovative Tool Has Become Routine. Arch Bronconeumol (Engl Ed). 2020 Apr;56(4):201-203. doi: 10.1016/j.arbres.2019.06.020. Epub 2019 Aug 3. No abstract available. English, Spanish. PMID 31383496
- [Background] Santana PV, Cardenas LZ, Albuquerque ALP, Carvalho CRR, Caruso P. Diaphragmatic ultrasound: a review of its methodological aspects and clinical uses. J Bras Pneumol. 2020 Nov 20;46(6):e20200064. doi: 10.36416/1806-3756/e20200064. eCollection 2020. PMID 33237154
- [Background] Boussuges A, Rives S, Finance J, Bregeon F. Assessment of diaphragmatic function by ultrasonography: Current approach and perspectives. World J Clin Cases. 2020 Jun 26;8(12):2408-2424. doi: 10.12998/wjcc.v8.i12.2408. PMID 32607319